CLINICAL TRIAL: NCT03044938
Title: Acute Effect of Salbutamol on Heart Rate and Blood Pressure During Exercise in Patients With Moderate or Severe Asthma and Healthy Subjects: Randomized, Double-blind, and Crossover Study
Brief Title: Acute Effect of Salbutamol on Heart Rate and Blood Pressure During Exercise in Patients With Moderate or Severe Asthma and Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Ibirapuera (Other)
Collaborators: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Felipe Augusto Rodrigues Mendes, Full Professor of Physiotherapy at the Ibirapuera University, Universidade Ibirapuera
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1.574.833
Record Dates: First submitted 2017-01-23; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Asthma; Heart Rate Fast
Keywords: Asthma; Salbutamol; Exercise; Heart Rate; Blood pressure
MeSH Terms: conditions — Asthma; Tachycardia; Motor Activity | interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: Randomized Clinical trial, controlled, double-blind and crossover
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salbutamol (Experimental): Salbutamol is a bronchodilator that relaxes the muscles of the airways and increases the flow of air to the lungs. With the aid of a spacer, 400mcg of the drug will be administered once during the protocol.
  Interventions: Drug: salbutamol
- Placebo (Placebo Comparator): Inoculant treatment through a substance that does not have an inherent power to produce an effect that is desired or expected. Four placebo puffs will be offered through a device similar to the salbutamol intervention device.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: salbutamol — Salbutamol or albuterol is a short-acting β2 adrenergic receptor agonist used for the relief of bronchospasm in conditions such as asthma and chronic obstructive pulmonary disease.
  Other Names: Albuterol
  Arms: Salbutamol
Drug: Placebo — Neutral preparation for pharmacological effects, given in substitution of a medicine, for the purpose of provoking or controlling reactions, ger. Of a psychological nature, accompanying such a therapeutic procedure.
  Other Names: Falso
  Arms: Placebo

SUMMARY:
Contextualization: Exercise is a common triggers of bronchospasm in patients with asthma and healthy subjects. To prevent these symptoms frequently they have to use Short-Acting Beta2-Agonists. However, the cardiovascular effects of salbutamol during and after exercise remain poorly known.

Objective: To evaluate the effect of salbutamol on heart rate and blood pressure during exercise in patients with moderate or severe asthma and healthy individuals.

Methods: A randomized, double-blind, crossover study will be conducted which 13 individuals with moderate or severe persistent asthma and 13 healthy individuals aged between 20 to 59 years.

Patients will perform a maximal effort test on 2 nonconsecutive days, with either 400mcg Salbutamol or 4 placebo puffs. The order of use of placebo or salbutamol will be drawn. During the protocol, heart rate, blood pressure, perception of exertion and peak expiratory flow will be monitored.

ELIGIBILITY:
Inclusion Criteria for asthmatics:

* Have the diagnosis of moderate or severe asthma according to the clinical criteria described in the literature
* Be between 20 and 59 years of age
* Being from the Asthma Assistance and Research Center (NAPA) of University of São Paulo Faculty of Medicine Clinics Hospital
* Have treatment at the outpatient clinic for at least 3 months,
* Have a stable clinical condition for at least 30 days
* Make use of the optimized medicine daily
* Read and signed the TCLE approved by the Ethics and Research Committee of the Ibirapuera University (UNIB) under opinion nº 1,574,833

Exclusion Criteria for asthmatics:

* Individuals diagnosed with another lung disease,
* Have psychiatric, musculoskeletal or cardiovascular diseases,
* Being smokers
* Being pregnant
* Practice regular physical activity.

Criterion for inclusion of healthy individuals

* Be between 20 and 59 years of age
* Healthy individuals
* Both genders
* Age between 20 and 59 years
* Read and signed the TCLE approved by the Ethics and Research Committee of the Ibirapuera University (UNIB) under opinion nº 1,574,833

Criteria for the exclusion of healthy individuals

* Pregnant women
* Smokers
* Psychic diseases
* Osteomuscular diseases
* Practitioners of regular exercise
* Physical Activity Readiness Questionnaire (PAR-Q)

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-08-06 (Actual); Primary Completion 2016-08-06 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
Heart rate | Baseline up to 1 hour and after 1 week.
  It is being considered that the asthmatic heart rate will increase after the use of salbutamol and that the increase will remain during and after the exercise, in relation to the placebo intervention. To evaluate this variable, the Polar RS800cx heart rate monitor will be used, where the participant will have his heart beats monitored beat to beat until the end of the protocol.

SECONDARY OUTCOMES:
Blood pressure | Baseline and for 1 hour and after 1 week again.
  It is being considered that the systemic arterial pressure (SBP) of the asthmatic will not have significant alteration after the use of salbutamol during and after the exercise. To evaluate this variable, a Solidor manual sphygmomanometer and a supermed stethoscope will be used. The SBP will be measured after 10 minutes of initial rest, 15 minutes after administration of the drug, every 3 minutes during the physical test and every 5 minutes for 20 minutes at rest.
Peak flow | Baseline, 15 minutes final and after 1 week.
  Due to improved airflow brought by the drug, the peak expiratory flow is expected to increase with the use of salbutamol.
Subjective perception of Borg | 1 hour and after 1 week .
  The modified borg subjective perception scale will be used, where the perception of effort will be reported by a scale ranging from 0 to 10. The scale will be applied during the stress test every 3 minutes and during the final rest phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Jaqueline Ribas de Melo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No